CLINICAL TRIAL: NCT04603716
Title: Effects of Concentric Versus Eccentric Muscle Energy Technique on Pain, Muscle Length and Function in Upper Cross Syndrome
Brief Title: Concentric Versus Eccentric Muscle Energy Technique on Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCRS/20/1010 Sadia Khalid
Record Dates: First submitted 2020-10-19; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Neck Syndrome
Keywords: upper cross syndrome,; MET,; NDI,; NPRS
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric Muscle Energy Technique (Experimental): conventional physical therapy Along with eccentric muscle energy technique
  Interventions: Other: Eccentric Muscle Energy Technique
- concentric muscle energy technique (Experimental): Conventional physical therapy along with concentric muscle energy technique
  Interventions: Other: Concentric muscle energy technique

INTERVENTIONS:
Other: Eccentric Muscle Energy Technique — Conventional Treatment given to both groups (Hot pack for 15 minutes, Mobilization, AROM Exercises 10 sets x 3days in a week)
  Reciprocal inhibition of target muscle (i.e. levator scapulae ,pectoralis major, upper trapezius) causing relaxation, patient force is minimal towards maximal therapist force, 5-7 repetition for 2-4seconds 3 days in a week up to 6 weeks.
  Muscle is taken from shortened to lengthened position.
  Arms: Eccentric Muscle Energy Technique
Other: Concentric muscle energy technique — Group B: Concentric Muscle Energy Technique: (Autogenic inhibition of target muscle (i.e. levator scapulae ,pectoralis major, upper trapezius) patient force is greater than therapist force, 5-7repitition for 3-4seconds)Muscle is taken from lengthened to shortened position.
  On eligible participants baseline assessment was done,3 session were given 3days per week, post intervention assessment was taken at 1st 3rd and 6th week
  Arms: concentric muscle energy technique

SUMMARY:
This project was a Randomized control trial conducted to check the effects of eccentric and concentric muscle energy techniques on patients with upper cross syndrome so that we can have best treatment option for patients with upper cross syndrome, duration was of 6months,convenient sampling was done, subject following eligibility criteria from Mansoura hospital female physiotherapy department, Lahore were randomly allocated in two groups via lottery method, baseline assessment was done, Group A participants were given conservative treatment along with eccentric muscle energy technique and Group B participants were given conservative treatment along with concentric muscle energy technique than on 1st,3rdand 6th week post intervention assessment was done via neck disability index, Numeric rating scale, inches tape method,3 sessions per week were given, data was analyzed by using SPSS version 26.

DETAILED DESCRIPTION:
In Upper cross syndrome upper trapezius, pectoralis major, and levator scapulae become tight and rhomboids , serratus anterior, middle and lower trapezius, and deep neck flexors, including scalene becomes weak. The postural muscles have tendency to become tight while the phasic muscles have tendency to become weak and inhibited. Thus typical pattern of altered posture and muscular imbalance occurs whenever dysfunction of muscle start. mainly muscular imbalance between weak and tonic muscles leads toward this upper cross syndrome. Soft tissue and cervical spine disorders are found out to be the major contributor in neck pain but when postural abnormality becomes the reason behind neck ache than this is categorized as Upper cross syndrome due to this imbalance in muscles our body has to suffer from severe consequences.rounded shoulder posture is a result of protracted girdle of shoulder due to muscular imbalances between agonist and antagonist muscles resulting in extreme pain and exaggerated cervical curvature.Imbalanced stress on cervical vertebrae is responsible in creating extra pull on neck and head similarly change in normal posture is responsible in overloading, weakening or tightening of cervical area. Characteristics of patient presenting with UCS will have forward head posture, kyphosis ,hunch of thoracic spine (rounded shoulder),winged scapulae, protracted and elevated shoulder and reduced thoracic spine mobility. UCS with the passage of time can detoriate persons physical fitness and health ,it is not only responsible for changes in posture of upper back i.e hypokyphosis over time, but it is also responsible for inducing respiratory problems including asthma. It also cause neck back shoulder and chest wall pain, this pain can be caused by muscular imbalance leading to overuse and fatigue of muscle because of movement dysfunction of back and neck.when muscles become fatigued they start generating more amount of inflammatory chemicals resulting in becoming more sore and increased spasticity. With the passage of time biomechanical and postural changing will induce osteoarthritis in upper thoracic and lower cervical spine in early ages. Functional Shoulder impingement syndrome is also considered to be another complication of Upper cross syndrome. Therefore it is necessary to correctly diagnose and treat this condition before its complication starts worsening.

ELIGIBILITY:
Inclusion Criteria:

* 6 month chronic neck pain
* upper cross syndrome:
* Clinical picture (Postural Changes):
* Forward head posture
* Increased cervical lordosis and thoracic kyphosis
* Elevated and protracted shoulders (Rounded shoulders)
* A hunched upper back
* Rotation or abduction and winging of the scapula

  * Test: Janda test: Patient supine tries to elevate the head from the couch. Normally the lordosis will disappear and the chin will touch the sternum. Otherwise pathological picture shows that the head is lifted with the very tense neck muscles

Exclusion Criteria:

* Patients having any serious trauma on neck i.e. whiplash injury
* Spinal fracture
* Cervicogenic headache
* History of systemic disease RA, SLE, TUMOR
* psychiatric disorder
* Any Red flag

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-12-30 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 6th Week
  10-item questionnaire that measures a patient's self-reported neck pain related disability. A higher NDI score means the greater a patient's perceived disability due to neck pain. 10 item score from 0-5.maximum score is 50.
  * 0 to 4(0-8%)=no disability
  * 5 to14(19-28%)=mild
  * 15 to24(30-48%)=moderate
  * 25 to 34 (50-64%)=severe
  * Above 34(70-80%)=complete.
    10-item questionnaire that measures a patient's self-reported neck pain related disability. A higher NDI score means the greater a patient's perceived disability due to neck pain. 10 item score from 0-5.maximum score is 50.
  * 0 to 4(0-8%)=no disability
  * 5 to14(19-28%)=mild
  * 15 to24(30-48%)=moderate
  * 25 to 34 (50-64%)=severe
  * Above 34(70-80%)=complete

SECONDARY OUTCOMES:
NPRS | 6th Week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain

OTHER OUTCOMES:
Inches Tape method | 6th Week
  Two bony landmarks were selected to measure the length of pectoralis major, upper trapezius, levator scapulae with the help of inches tape ,idea was taken from the Joint range of motion and muscle length testing-E-book by NB Reese,WD Bandy - 2016 - Elsevier Health Sciences

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur-Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Mansoora hospital, Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joshi S, Srivastava N. To Compare the Effectiveness of Active Release Technique and Conventional Physical Therapy in the Management of Upper Cross Syndrome. Indian Journal of Physiotherapy & Occupational Therapy. 2018;12(4).
- [Background] Rivera CE. Core and Lumbopelvic Stabilization in Runners. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):319-37. doi: 10.1016/j.pmr.2015.09.003. PMID 26616187
- [Background] Rajalaxmi V, Paul J, Nithya M, Lekha SC, Likitha B. Effectiveness of three dimensional approach of schroth method and yoga on pulmonary function test and posture in upper crossed syndrome with neck Pain-A double blinded study. Research Journal of Pharmacy and Technology. 2018;11(5):1835-9.
- [Background] Izzo R, Popolizio T, D'Aprile P, Muto M. Spinal pain. Eur J Radiol. 2015 May;84(5):746-56. doi: 10.1016/j.ejrad.2015.01.018. Epub 2015 Feb 13. PMID 25824642
- [Background] Yoo K-T, Lee H-S. Effects of therapeutic exercise on posture, pain and asymmetric muscle activity in a patient with forward head posture: Case report. Journal of Korean Society of Physical Medicine. 2016;11(1):71-82.
- [Background] Rajalaxmi V, Ranjani V, Paul J, Subramanian S, Cyrus BE, Pavithralochani V. Efficacy of Neck Stabilization and Postural Correction Exercise on Pain, Posture, Disability, Respiratory Dysfuntions and Mental Status in Desk Job Workers-A Randomised Controlled Double Blinded Study. Research Journal of Pharmacy and Technology. 2019;12(5):2333-8.
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Mujawar JC, Sagar JH. Prevalence of Upper Cross Syndrome in Laundry Workers. Indian J Occup Environ Med. 2019 Jan-Apr;23(1):54-56. doi: 10.4103/ijoem.IJOEM_169_18. PMID 31040591
- [Background] Tiefel K. The Efficacy of Treatment for Upper Crossed Syndrome and the Involvement of Chiropractic. 2012.
- [Background] Shahzad AN, Shakil-ur-Rehman S, Rafique N. Effectiveness of eccentric and concentric muscle energy techniques on hamstring length in healthy population. Rawal Medical Journal. 2019;44(2):350-2.
- [Background] Osama M, Tassadaq N, Malik RJ. Effect of muscle energy techniques and facet joint mobilization on spinal curvature in patients with mechanical neck pain: A pilot study. J Pak Med Assoc. 2020 Feb;70(2):344-347. doi: 10.5455/JPMA.14189. PMID 32063632
- [Background] Osama M, Shakil Ur Rehman S. Effects of static stretching as compared to autogenic inhibition and reciprocal inhibition muscle energy techniques in the management of mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 May;70(5):786-790. doi: 10.5455/JPMA.9596. PMID 32400728
- [Background] Rana AA, Ahmad A, Gillani SA, Idrees MQ, Awan I. Effects of conventional physical therapy with and without muscle energy techniques for treatment of Upper Cross Syndrome. Rawal Medical Journal. 2020;45(1):127-32.
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028
- [Background] Reese NB, Bandy WD. Joint range of motion and muscle length testing-E-book: Elsevier Health Sciences; 2016.